CLINICAL TRIAL: NCT04544722
Title: Clinical Study of Jianfei Kangfu Cao in the Treatment of Primary Sjogren's Syndrome Associated Interstitial Lung Disease.
Brief Title: Clinical Study of Jianfei Kangfu Cao in the Treatment of pSS-ILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jianfei Kangfu Cao
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-08

CONDITIONS: Primary Sjogren's Syndrome; Interstitial Lung Disease
Keywords: Safety; Efficacy; Primary Sjogren's syndrome; Interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jianfei Kangfu Cao (Experimental): The original treatment and Jianfei Kangfu Cao, once a day, 30 minutes each time.
  Interventions: Behavioral: Jianfei Kangfu Cao
- Lung rehabilitation training (Active Comparator): The original treatment and the lung rehabilitation training, once a day, 30 minutes each time.
  Interventions: Behavioral: lung rehabilitation training

INTERVENTIONS:
Behavioral: Jianfei Kangfu Cao — The original treatment and Jianfei Kangfu Cao, once a day, 30 minutes each time.
  Arms: Jianfei Kangfu Cao
Behavioral: lung rehabilitation training — The original treatment and the lung rehabilitation training, once a day, 30 minutes each time.
  Arms: Lung rehabilitation training

SUMMARY:
This study will evaluate the safety and efficacy of Jianfei Kangfu Cao in the treatment of primary Sjogren's syndrome associated interstitial lung disease.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, positive control clinical trial with a course of 24 weeks.

1. Random scheme:the DAS for Interactive Web Response System(IWRS) will be used to calculate and distribute random numbers and dispensing drugs.
2. Blind method ：The test process will be in a double-blind state.
3. Control drug: The lung rehabilitation training will be used as control in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. According to the 2012 ACR classification of primary Sjogren's syndrome .
2. CT confirmed interstitial lung disease;
3. DLCO≧40%;
4. Stable treatment for at least 12 weeks;
5. Patients with good compliance should sign informed consent before the tria.

Exclusion Criteria:

1. The patient is using or has used anti pulmonary fibrosis drugs;
2. Pulmonary infection, tumor and other connective tissue diseases;
3. Chronic obstructive pulmonary disease, bronchial asthma and tuberculosis;
4. Patients with severe hypertension, diabetes and heart, liver and renal failure;
5. Women with reproductive needs;
6. Idiopathic pulmonary interstitial disease;
7. The researcher thinks that it is not suitable to participate in this experiment;
8. Participants in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
FVC | 24 weeks
  FVC is an index of lung function.
CAT score | 24 weeks
  Cat questionnaire includes eight questions, the core of which is cough, expectoration, chest tightness, sleep, energy, emotion, and two tolerance evaluation indexes, namely, exercise endurance and daily exercise influence. According to the patient's own situation, each item was scored accordingly (0-5), and the cat score range was 0-40

SECONDARY OUTCOMES:
6MWD | 24 weeks
  Six minutes walk test is a kind of exercise test for the functional state of patients with moderate and severe cardiopulmonary disease.
ESSDAI | 24 weeks
  Evaluation of Sjogren's disease activity
ESSPRI | 24 weeks
  EULAR SS Patient Reported Index

CONTACTS AND LOCATIONS:
Overall Officials: Zhujing Zhu, Ph.D, Principal Investigator — Longhua Hospital; Jianchun Mao, Master, Study Chair — Longhua Hospital; Huanru Qu, Ph.D, Study Chair — Longhua Hospital
Locations (1):
- Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No